CLINICAL TRIAL: NCT04838769
Title: Water Vapor Thermotherapy vs. Combination Pharmacotherapy for Symptomatic Benign Prostatic Hyperplasia Refractory to Alpha Blocker Monotherapy in Sexually Active Men: A Multicenter Randomized Controlled Trial
Brief Title: REZŪM vs. Dual Drug Therapy for Symptomatic Benign Prostatic Hyperplasia in Sexually Active Men
Acronym: VAPEUR
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: U0693
Record Dates: First submitted 2021-04-06; First posted 2021-04-09 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Benign Prostatic Hyperplasia (BPH)
Keywords: Prostate; REZŪM; Water vapor thermotherapy; Lower urinary tract symptoms; BPH; LUTS
MeSH Terms: conditions — Prostatic Hyperplasia; Lower Urinary Tract Symptoms | interventions — Adrenergic alpha-Antagonists; 5-alpha Reductase Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- REZŪM (Active Comparator): Subjects randomized to receive the REZŪM treatment will receive standardized treatment, following the Instruction for Use (IFU). The REZŪM System is intended to relieve symptoms, obstructions, and reduce prostate tissue associated with benign prostatic hyperplasia (BPH). It is indicated for men with a prostate volume ≥ 30 ml. The REZŪM System is also indicated for treatment of prostate with hyperplasia of the central zone and/or a median lobe.
  1:1 randomization will occur via the electronic data capture (EDC) system.
  Interventions: Device: REZŪM
- Dual Drug Therapy (Active Comparator): Subjects assigned to dual drug therapy will be treated with the local formulary preferred choice of commercially available urinary selective alpha blocker and 5-alpha reductase inhibitor. This arm will therefore represent local standard of care.
  Interventions: Drug: alpha blocker and 5-alpha reductase inhibitor

INTERVENTIONS:
Device: REZŪM — Subjects randomized to receive the REZŪM treatment will receive standardized treatment, following the Instruction for Use.
  Arms: REZŪM
Drug: alpha blocker and 5-alpha reductase inhibitor — Subjects assigned to dual drug therapy will be treated with the local formulary preferred choice of commercially available urinary selective alpha blocker and 5-alpha reductase inhibitor. This arm will therefore represent local standard of care.
  Other Names: Dual Drug Therapy
  Arms: Dual Drug Therapy

SUMMARY:
The study objective is to compare water vapor thermotherapy with the REZŪM™ System to dual drug therapy for the treatment of symptomatic benign prostatic hyperplasia refractory to alpha-blocker monotherapy in sexually active men.

DETAILED DESCRIPTION:
STUDY OBJECTIVE - To compare water vapor thermotherapy with the REZŪM™ System to dual drug therapy for the treatment of symptomatic benign prostatic hyperplasia refractory to alpha-blocker monotherapy in sexually active men.

STUDY DESIGN - Multicenter open-label randomized controlled parallel-group post-market trial.

STUDY TREATMENTS AND RANDOMIZATION - Subjects will be randomly assigned to REZŪM or dual drug therapy treatments; 1:1 randomization via the electronic data capture (EDC) system. Both treatments are commercially available. Subjects randomized to receive the REZŪM treatment will receive standardized treatment and subjects randomized to dual drug therapy will receive the local formulary preferred choice of urinary selective alpha blocker and 5-alpha reductase inhibitor.

VISIT SCHEDULE - Study visits are at: enrollment/baseline, treatment, 3 months, 6 months, and yearly follow-up through 2 years.

ELIGIBILITY:
Inclusion Criteria:

1. Sexually active male subjects ≥ 45 years of age who have persistent non-neurogenic lower urinary tract symptoms refractory to first-line treatment with single agent Alpha Adrenoceptor Antagonist therapy
2. Subject is willing and able to answer all domains of MSHQ
3. Completed IPSS questionnaire with score ≥ 13 within 6 months prior to enrollment
4. Peak urinary flow rate (Qmax): ≤ 15 ml/sec with minimum voided volume of ≥ 150 ml within 6 months prior to enrollment
5. Post-void residual (PVR) ≤250 ml within 6 months prior to enrollment
6. Prostate volume ≥ 30 ml as measured by transrectal ultrasound or Magnetic Resonance Imaging within 3 months prior to enrollment
7. Subject is willing and capable of providing informed consent
8. Subject is willing and capable of participating in all visits associated with this study at an approved clinical study site and at the intervals defined by this Clinical Investigational Plan (CIP)
9. France subjects only: subjects must be affiliated to national security insurance

Exclusion Criteria:

1. Inability to participate in full duration of study
2. Prior surgical treatment for BPH
3. Increased risk of bleeding
4. Presence of Genitourinary Cancer or other pelvic cancer
5. Functional issues with bladder
6. Presence of active infection in genitourinary tract
7. Structural and Anatomic issues with urinary tract and renal function
8. Concomitant Drug Therapy
9. Temporal restraints and risks for general anaesthesia or comorbidity that would elevate risk of participation

Min Age: 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Sexually active male subjects
Enrollment: 154 (Actual)
Dates: Start 2021-09-15 (Actual); Primary Completion 2025-12-11 (Actual); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
International Prostate Symptom Score (IPSS) change | From Baseline to 12 months
  Primary Statistical Hypothesis: Change in IPSS score will be compared between groups. IPSS score ranges from 0 to 35 with higher scores indicating worse symptoms.
Male Sexual Health Questionnaire (MSHQ) total score change | From Baseline to 12 months
  Change in MHSQ score will be compared between groups. MHSQ score ranges from 0 to 125 with higher scores indicating better outcomes.

SECONDARY OUTCOMES:
Disease Progression | End of available follow-up, up to 24 months
  Disease progression, defined as occurrence of any of the following:
  * Surgical retreatment for LUTS/BPH
  * Urinary retention requiring urinary catheterization after 90 days post-treatment
  * IPSS increase from baseline by ≥ 4 points
  * Introduction of a new drug agent to treat LUTS/BPH

CONTACTS AND LOCATIONS:
Overall Officials: Romain Mathieu, Professor, Principal Investigator — CHU Rennes, Hôpital Pontchaillou; Evanguelos Xylinas, Ass. Prof., Principal Investigator — Hôpital Bichat
Locations (21):
- Australia (2):
  - Epworth Healthcare, Melbourne
  - Australian Clinical Trials, Wahroonga
- France (19):
  - Centre Hospitalier du Pays d'Aix, Aix-en-Provence
  - CHU d'Angers, Angers
  - CHU de Bordeaux, Bordeaux
  - CHU Grenoble, Grenoble
  - Centre Hospitalier Universitaire de Lille, Lille
  - Hôpital Privé La Louvière, Lille
  - Hospices Civils de Lyon, Lyon
  - CHU de Nice, Nice
  - Hôpital Bichat, Paris
  - Hôpital Cochin, Paris
  - Institut Mutualiste Montsouris, Paris
  - Hôpital privé Francheville, Périgueux
  - Clinique La Croix du Sud, Quint-Fonsegrives
  - CHU de Rennes, Rennes
  - CHU de Rouen, Rouen
  - Clinique Saint Hilaire, Rouen
  - Centre Hospitalier Privé Saint Grégoire, Saint-Grégoire
  - CHU de Toulouse, Toulouse
  - Clinique Pasteur, Toulouse

IPD SHARING:
Plan to Share IPD: No